CLINICAL TRIAL: NCT04943822
Title: Kaohsiung Chang Gung Memorial Hospital Nursing Department
Brief Title: The Effectiveness of APP Intervention on Home Self-care Ability and Quality of Life of Patients With Intestinal Stoma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: fung
Record Dates: First submitted 2021-06-09; First posted 2021-06-29 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2022-06

CONDITIONS: Quality of Life; Mobile Apps; Ostomy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional education service program (Placebo Comparator): Including the written and verbal health education on preoperative preparation, stoma surgery and postoperative stoma care. At discharge, ET nurses offered teaching information and support for patients, including selection of pouching appliances, drug instructions, health education At each outpatient follow-up, both stomas and patients needed to be assessed. The condition of stoma and peristomal skin, nature and volume of effluent, date of pouch appliances and stoma complications were recorded by ET nurses.
  Interventions: Other: A new APP
- mobile care device (Experimental): The participants in the intervention group were given the same routine care as the control group pre- and postoperatively. ET nurses taught patients and their family members how to use the home care mobile app before discharge. The home care mobile app was designed and developed for the discharged stoma patients by the research team and an information technology company in March 2021. Patients could receive stoma care from ET nurses through this mobile app at home, not just going to an outpatient clinic. The Major function modules of this mobile app were as follows: (a) appointment: The app users were able to complete the basic personal and medical information and make an appointment with the ET nurse; (b) photograph diagnosis: The ET nurses could make a diagnosis based on the patients' uploaded stoma photographs; and (c) consultation: Patients were able to contact their ET nurses for help and support. This mobile app was used to supplement the outpatient follow-up.
  Interventions: Other: A new APP

INTERVENTIONS:
Other: A new APP — A new APP for prevention and treatment of complications of intestinal peristomal skin

SUMMARY:
Colorectal cancer is the third leading cause of cancer-related deaths in Taiwan.

In the United States, colorectal cancer is the third most common cancer diagnosis and mortality.

According to the databases of the Bureau of National Health Insurance (BNHI), in 2003-2006, a total of 15,805 patients with colorectal surgery were included, and 27.11% were treated with ostomy, while 90.45% were colostomy and 9.55% were ileostomy.

The domestic and foreign researches related to enterostomy mostly use cross-sectional research methods. The quality of life, knowledge of self-care and self-care needs of different postoperative methods of colorectal cancer have not been specifically improved for patients with enterostomy. The research on self-care ability and quality of life is for reference. In other countries, enterostomy care has gradually moved from medical institutions to community care, but community nurses generally have no relevant care skills. Advances in mobile technology such as smartphones and other mobile applications have created more opportunities for individuals to receive health-related treatments, anytime, anywhere and anywhere. In the United States, 93% of adult gastroenterology patients have smartphones in medical teaching hospitals, and most of them are interested in using health-related applications. In addition, previous studies have shown the potential benefits and efficacy of mobile devices for self-care patients in diabetes, obesity and cancer. However, there are limited studies on the feasibility and effectiveness of mobile applications for enterostomy care. Researchers want to explore the effectiveness of mobile device intervention on home self-care ability and quality of life of patients with intestinal stoma.

DETAILED DESCRIPTION:
1. Background and research purpose Colorectal cancer has been ranked first in the nation's cancer incidence for 11 consecutive years. Clinically, the surgical treatment of rectal cancer is more difficult than that of colorectal cancer. On the one hand, it is the anatomical location factor. Unlike colorectal cancer, which is located in the abdominal cavity, rectal cancer is located in the narrower pelvic cavity with many bones surrounding it. In particular, the pelvic cavity of men is smaller than that of women, so the space available for surgery is relatively smaller than that of the large intestine. Cancer is much less. On the other hand is the consideration of preserving the anus. When removing a tumor that grows in the colon, there is basically no question of whether to preserve the anus or not, because the large intestine is very long. However, in order to clean the tumor, the doctor will leave a certain safe distance between the front and rear ends of the tumor, that is, an extra 5-10 cm of cut. However, for rectal tumors, most clinically patients want to preserve the anus. Therefore, the current safe distance from the end of the tumor during rectal cancer resection is best to exceed 1 cm.

   Therefore, for patients with rectal cancer, the way of defecation will definitely change after surgery, but the impact will be large or small. It is generally recommended to adjust the diet, such as reducing the intake of fiber such as fruits and vegetables to reduce bowel movements. Some patients think that the uncertainty of dietary restrictions and defecation will affect the quality of life, and they choose permanent artificial anus. Although patients with colorectal cancer usually do not need to remove the anus, they sometimes need temporary artificial anus, such as obstructive colorectal cancer. , First do a temporary artificial anus to help defecation, the purpose is to reduce pressure, let the swollen belly disappear, and then perform surgery to remove the tumor and remove the artificial anus. Although this artificial anus is only temporary, it is not permanent. Among them, about 21% to 70% of enterostomy patients will have some types of complications. These complications are related to stoma dysfunction, insufficient stoma positioning and poor self-care ability. It may cause dermatitis, bleeding, prolapse, necrosis, hernia, edema, waste including leakage, tracheal hernia, stenosis and retraction. Nowadays, advances in mobile technology, such as mobile applications such as smartphones, have created more opportunities for individuals to treat health-related treatments, anytime, anywhere.
2. Research motivation The use of apps as a tool for teaching, nursing and diagnosing skin lesions is a very innovative tool that allows learners to generate interest and motivation to learn more, because the use of apps on mobile devices in the health care sector is higher than that of books. Out of 45%-85%. The purpose of this study is to investigate the effectiveness of using mobile devices to intervene in the self-care ability and quality of life of patients with intestinal stoma.
3. Research design and objects A single blind-experimental design is adopted. First, those who meet the acceptance criteria and are willing to participate in the research are selected and assigned to the experimental and control groups by random assignment by the computer random number table. It is estimated that 2 people will be needed Nursing staff were admitted in the rectal anal treatment room. Participants were randomly assigned to receive routine discharge care and mobile device guidance or routine outpatient follow-up. Data were collected before the patient was discharged, 1 month, 2 months and 4 months after discharge . The structured questionnaire is filled in by the patient or the researcher.
4. statistical methods Descriptive statistics, including frequency distribution and percentage, average and standard deviation, median and interquartile range, and other data to describe the distribution of data; first use the Kolmogorov-Smirnov test to determine whether the data conform to normality Distribution; univariate analysis adopts independent-sample t test or Mann-Whitney U test to compare the difference between the experimental group and the control group in the continuous variables collected, Chi-square test (chi-square test) or Fisher's exact test (Fisher's exact test) compares the difference between the categorical variables collected in the experimental group and the control group; further, binary logistic regression and stepwise regression are used. Regression screening mode method is used to analyze multiple variables to find out the important explanatory factors related to the involvement of mobile devices in personal attributes, self-care ability and quality of life.

ELIGIBILITY:
Inclusion Criteria:

1. diagnosed with primary colorectal cancer;
2. at least 20 years of age;
3. able to read and speak Mandarin;
4. own a smartphone and willingness to use the mobile app after discharge The exclusion criteria

1.having other types of cancer; 2.having visual, hearing and/or cognitive impairments/mental disorders; 3.alcohol or drug abuse; 4.dying or having any surgical complications.

Ages: 20 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Quality of life improvement | One and a half years
  The Enterostomy- QOL was comprised of 30 questionnaires, it covered seven domains: relations with family and friends, Sleep, activity, sexual activity, social relationship, physiology and psychology. The responses rated on a4-point scale Likert scale (1: extremely, 2: quite a lot, 3: somewhat, 4: not at all). The possible scores range was from 37 to 148. Higher scores indicated that patient had a higher level of quality of life.

SECONDARY OUTCOMES:
Self-care ability improvement | One and a half years
  Assessment scale of self-care ability of enterostomy care was a quantitative scale for nursing staff to evaluate self-care skills in patients with enterostomy. It consisted of 7 items related to: Prepare items, removing the pouching system, measuring the enterostomy diameter, adjusting the size of the enterostomy diameter in a new stoma appliance, skin care, fitting a new enterostomy appliance, and emptying procedure. Each skill was rated on a 4-point scale: Likert scale (1: not at all, 2: some, 3: quite a lot, 4: very much).
hospital medical record for clinical data | One and a half years
  Clinical data including disease, stoma site and type were collected from hospital medical records.
Stoma complications | One and a half years
  It contained mucocutaneous separation, stoma necrosis, peristomal dermatitis, retraction, prolapsed, stenosis and parastomal hernia

CONTACTS AND LOCATIONS:
Locations (1):
- Hsing Fang Ko, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No